CLINICAL TRIAL: NCT02333929
Title: Validation of Rivaroxaban Assay for US Registration
Status: Completed | Type: Observational
Sponsor: Diagnostica Stago (Industry)
Responsible Party: Sponsor
Other Study IDs: VSP P391-US
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Patients Receiving Rivaroxaban Treatment
Keywords: rivaroxaban; NOAC; anti-Xa activity; method comparison; LCMS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- VTE prevention: Prophylaxis of VTE in patients undergoing knee or hip replacement surgery (10 mg OD): orthopaedic department of the hospital will be in charge of the sample collection.
  Interventions: Device: STA- Rivaroxaban Calibrator&Control
- DVT/PE treatment: Treatment of deep vein thrombosis (DVT), pulmonary embolism (PE), and risk reduction of DVT and PE recurrence; (15 mg BID for 3 weeks then 20 mg OD): different departments of the hospital will be in charge of the sample collection (samples can come e.g., from emergency room, vascular lab or cancer unit).
  Interventions: Device: STA- Rivaroxaban Calibrator&Control
- SPAF: Stroke prevention and reduction of systemic embolism in non-valvular patients with atrial fibrillation (SPAF) (20 mg OD): cardiology department of the hospital will be in charge of the sample collection.
  Interventions: Device: STA- Rivaroxaban Calibrator&Control

INTERVENTIONS:
Device: STA- Rivaroxaban Calibrator&Control — One sample blood collected per patient the day of the treatment (drawn soon after the the drug intake)

SUMMARY:
The objective of the study is to demonstrate the performances of the STA® - Rivaroxaban Calibrator and STA® - Rivaroxaban Control in combination with the STA® - Liquid Anti-Xa to determine the quantity of rivaroxaban in plasma samples by measurement of its direct anti-Xa activity.

DETAILED DESCRIPTION:
The study is a method comparison between a reference method (LCMS) and the candidate device.

Between 90 and 120 samples obtained from patients treated by rivaroxaban will be collected on 3 sites in the US according to the inclusion and exclusion criteria detailed in the protocol. These samples will be frozen after the collection and sent to the hemostasis laboratories for testing and to a LCMS central laboratory validated for rivaroxaban measurement.

Results expressed in ng/mL obtained with STA® - Liquid Anti-Xa, used in combination with STA® - Rivaroxaban Calibrator and STA® - Rivaroxaban Control will be compared to the result obtained by the LCMS laboratory.

Diagnostica Stago will analyse the results thanks to regressions according to CLSI EP9-A3 recommendations (guideline dedicated to method comparison for quantitative assay) in order to support the equivalence between the 2 methods.

ELIGIBILITY:
Inclusion Criteria:

Between 30 and 40 samples/site obtained from patients treated with rivaroxaban.(ideally 10-15 samples per indication and per site depending on the site practices):

* Prophylaxis of VTE in patients undergoing knee or hip replacement surgery (10 mg OD): orthopaedic department of the hospital will be in charge of the sample collection.
* Treatment of deep vein thrombosis (DVT), pulmonary embolism (PE), and risk reduction of DVT and PE recurrence; (15 mg BID for 3 weeks then 20 mg OD): different departments of the hospital will be in charge of the sample collection (samples can come e.g., from emergency room, vascular lab or cancer unit).
* Stroke prevention and reduction of systemic embolism in non-valvular patients with atrial fibrillation (SPAF) (20 mg OD): cardiology department of the hospital will be in charge of the sample collection.

Exclusion Criteria:

* Patients less than 18 years old
* Patients under other anti-coagulant treatment
* Samples that are not collected, stored, or handled in accordance with sample collection procedures defined in CLSI H21-A5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving rivaroxaban treatment for one of the 3 drug indications cleared in the US
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of participants tested once during their rivaroxaban treatment | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: James Groce, Pharm D., Principal Investigator — Cone Health
Locations (1):
- Lehigh Valley Health Nrwork, Allentown, Pennsylvania, United States

REFERENCES:
- [Background] Baglin T, Hillarp A, Tripodi A, Elalamy I, Buller H, Ageno W. Measuring Oral Direct Inhibitors (ODIs) of thrombin and factor Xa: A recommendation from the Subcommittee on Control of Anticoagulation of the Scientific and Standardisation Committee of the International Society on Thrombosis and Haemostasis. J Thromb Haemost. 2013 Jan 24. doi: 10.1111/jth.12149. Online ahead of print. PMID 23347120
- [Background] Favaloro EJ, Lippi G. The new oral anticoagulants and the future of haemostasis laboratory testing. Biochem Med (Zagreb). 2012;22(3):329-41. doi: 10.11613/bm.2012.035. PMID 23092064